CLINICAL TRIAL: NCT04402190
Title: Hypotonic Hyponatremia: Criteria for the Correct Classification of Its Etiology and of Patient Volume Status at the Access in the Emergency Department and at the Subsequent Re-evaluation in Hospital Wards
Brief Title: Hypotonic Hyponatremia: Criteria for the Correct Classification of Its Etiology and of Patient Volume Status
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Ezio Ghigo, Medical Doctor, Full Professor in Endocrinology, A.O.U. Città della Salute e della Scienza
Other Study IDs: IPSO-URG
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Hyponatremia; Hyponatremia With Extracellular Fluid Depletion; Hyponatremia With Normal Extracellular Fluid Volume; Hyponatremia With Excess Extracellular Fluid Volume
Keywords: Hyponatremia; Hyponatremia with Extracellular Fluid Depletion; Hyponatremia with Normal Extracellular Fluid Volume; Hyponatremia with Excess Extracellular Fluid Volume; Hypotonic Hyponatremia; Volume Status; Intravascular Volume Status; Extracellular Fluid Volume Status; Copeptin
MeSH Terms: conditions — Hyponatremia; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hyponatremia is the most frequent electrolyte disorder encountered in clinical practice. The patient approach, however, is still problematic, above all because hyponatremia is a manifestation correlated to various pathological conditions, with complex etiopathogenesis.

Even though some algorithms have been proposed to correctly assess hyponatremia subtype classification and patient volume status, there is no single parameter that has proven to be able alone to perfectly achieve this result.

DETAILED DESCRIPTION:
Hyponatremia is the most frequent electrolyte disorder encountered in clinical practice and is often associated with increased mortality, morbidity and risk of hospitalization. The patient approach, however, is still problematic, above all because hyponatremia is a manifestation correlated to various pathological conditions, with complex etiopathogenesis.

The most commonly used classification of hypotonic hyponatremia is, nowadays, the one described in a famous review by Kumar and Berl (see Bibliography). Probably the most crucial point in this classification is represented by the correct assessment of Extracellular Fluid Volume Status (i.e. hypovolemia, euvolemia, hypervolemia).

Even though some algorithms have been proposed to correctly assess hyponatremia subtype classification and patient volume status, there is no single parameter that has proven to be able alone to perfectly achieve this result.

In the current study, the reference test (gold standard) for the definitive assessment of hyponatremia subtype classification and patient volume status was a post-discharge re-evaluation of all the available evidence (with the exception of plasma copeptin levels) carried out by two independent neuroendocrinologists with specific expertise in sodium disorders. In case of disagreement, the experts proceeded to a discussion and comparison of their opinions, in order to produce a shared one.

Using this gold standard, the main aims of this observational prospective study were:

1. to estimate the diagnostic accuracy of the clinicians in identifying the subtype of hyponatremia at the first evaluation of the patients in the ED and then at the admission to the wards;
2. to evaluate the diagnostic accuracy of the most important methods suggested by the literature (clinical, imaging, biochemical) for the assessment of Extracellular Fluid Volume.

In addition to this, in recent years copeptin has been shown to be a promising parameter for the evaluation of sodium disorders and water imbalances, but its diagnostic role in the setting of hyponatremic patients is still largely unknown. Therefore, a secondary objective of the study was to specifically evaluate the utility of copeptin (whose values - as specified before - were hidden to the neuroendocrinologists in charge of defining the gold standard diagnoses for each patient) for the assessment of hyponatremia subtype classification and patient volume status.

ELIGIBILITY:
Inclusion Criteria:

* Access to the emergency department (ED) of our hospital from Monday to Thursday, between 8 am and 6 pm (time constraint needed so that all the necessary laboratory analyzes could be correctly completed)
* Detection at the time of ED access of moderate-severe hyponatremia, defined as serum sodium < 130 mmol/L at blood gas analysis (BGA)
* Need for hospitalization

Exclusion Criteria:

* Programmed hospitalization that did not include access through the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted at the emergency department (ED) of our hospital in the time frames specified in the inclusion criteria with a detection, at the time of ED access, of moderate-severe hyponatremia (defined as serum sodium < 130 mmol/L at blood gas analysis).
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Subtype classification of hypotonic hyponatremia according to the overall judgment of the clinical case by the point-of-care clinician | At ED admission
  The point-of-care clinician was asked to provide a subtype classification of hypotonic hyponatremia according to his/her overall judgment of the clinical case (using Kumar and Berl classification classes as a reference frame). This will be compared to the gold standard reference (as defined in the "Study Description" Section). The strength of agreement (by Cohen's kappa) and the accuracy will thus be evaluated.
Subtype classification of hypotonic hyponatremia according to the overall judgment of the clinical case by the point-of-care clinician | At hospital ward admission
  The point-of-care clinician was asked to provide a subtype classification of hypotonic hyponatremia according to his/her overall judgment of the clinical case (using Kumar and Berl classification classes as a reference frame). This will be compared to the gold standard reference (as defined in the "Study Description" Section). The strength of agreement (by Cohen's kappa) and the accuracy will thus be evaluated.
Physical Examination (PE) as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Elements of PE relevant for ECF Volume Status assessment were recorded (blood pressure, heart rate, pulmonary crepitations/rales, jugular vein distension, peripheral edema, dry mucous membranes). The overall evaluation of ECF Volume Status based on PE alone will be compared to the gold standard reference (as defined in the "Study Description" Section).
Physical Examination (PE) as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Elements of PE relevant for ECF Volume Status assessment were recorded (blood pressure, heart rate, pulmonary crepitations/rales, jugular vein distension, peripheral edema, dry mucous membranes). The overall evaluation of ECF Volume Status based on PE alone will be compared to the gold standard reference (as defined in the "Study Description" Section).
Inferior Vena Cava (IVC) ultrasound evaluation as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  IVC diameter and collapsibility were recorded. The overall evaluation of ECF Volume Status based on IVC ultrasound evaluation alone will be compared to the gold standard reference (as defined in the "Study Description" Section).
Inferior Vena Cava (IVC) ultrasound evaluation as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  IVC diameter and collapsibility were recorded. The overall evaluation of ECF Volume Status based on IVC ultrasound evaluation alone will be compared to the gold standard reference (as defined in the "Study Description" Section).
Serum creatinine as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Serum creatinine (mg/dl) will be used to estimate GFR (ml/min) according to CKD-EPI formula. eGFR will then be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Serum urea as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Serum urea (mg/dl) will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Serum urea / serum creatinine ratio as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Serum urea / serum creatinine ratio will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Urine sodium as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Urine sodium (mmol/L), evaluated on a spot sample, will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Urine sodium / urine osmolality ratio as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Urine sodium / urine osmolality ratio will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Urine sodium / plasma osmolality ratio as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Urine sodium / plasma osmolality ratio will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Serum NT-proBNP as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Serum NT-proBNP (pg/ml) will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Serum NT-proBNP / urine sodium ratio as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Serum NT-proBNP / urine sodium ratio will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Serum creatinine as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Serum creatinine (mg/dl) will be used to estimate GFR (ml/min) according to CKD-EPI formula. eGFR will then be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Serum urea as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Serum urea (mg/dl) will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Serum urea / serum creatinine ratio as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Serum urea / serum creatinine ratio will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Urine sodium as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Urine sodium (mmol/L), evaluated on a spot sample, will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Urine sodium / urine osmolality ratio as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Urine sodium / urine osmolality ratio will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Urine sodium / plasma osmolality ratio as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Urine sodium / plasma osmolality ratio will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Plasma renin activity (PRA) as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  PRA (ng/ml/h) will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Uric acid as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Uric acid (mg/dl) will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.

SECONDARY OUTCOMES:
Plasma copeptin as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Plasma copeptin (pmol/L) will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Plasma copeptin / urine sodium ratio as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At ED admission
  Plasma copeptin / urine sodium ratio will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Plasma copeptin as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Plasma copeptin (pmol/L) will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.
Plasma copeptin / urine sodium ratio as a tool for the assessment of Extra-Cellular Fluid (ECF) Volume Status | At hospital ward admission
  Plasma copeptin / urine sodium ratio will be compared between three main groups of interest (i.e. hypovolemic, euvolemic and hypervolemic patients). As already previously described, these groups will be identified by the gold standard reference defined in the "Study Description" Section.

OTHER OUTCOMES:
Length of hospitalization | Up to 6 months after ED admission
  The length of hospitalization will be compared across subgroups according to hyponatremia subtype classification. As already previously described, these subgroups will be identified by the gold standard reference defined in the "Study Description" Section.
Overall mortality | Up to 6 months after ED admission
  All deaths occurring during hospitalization and/or within 6 months after hospital discharge will be registered. The overall mortality will be compared across subgroups (using a survival analysis model) according to hyponatremia subtype classification. As already previously described, these subgroups will be identified by the gold standard reference defined in the "Study Description" Section.

CONTACTS AND LOCATIONS:
Overall Officials: Ezio Ghigo, MD, Principal Investigator — AOU Città della Salute e della Scienza Torino
Locations (1):
- AOU Città della Salute e della Scienza, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spasovski G, Vanholder R, Allolio B, Annane D, Ball S, Bichet D, Decaux G, Fenske W, Hoorn EJ, Ichai C, Joannidis M, Soupart A, Zietse R, Haller M, van der Veer S, Van Biesen W, Nagler E; Hyponatraemia Guideline Development Group. Clinical practice guideline on diagnosis and treatment of hyponatraemia. Eur J Endocrinol. 2014 Feb 25;170(3):G1-47. doi: 10.1530/EJE-13-1020. Print 2014 Mar. PMID 24569125
- [Background] Fenske W, Maier SK, Blechschmidt A, Allolio B, Stork S. Utility and limitations of the traditional diagnostic approach to hyponatremia: a diagnostic study. Am J Med. 2010 Jul;123(7):652-7. doi: 10.1016/j.amjmed.2010.01.013. PMID 20609688
- [Background] Fenske W, Stork S, Blechschmidt A, Maier SG, Morgenthaler NG, Allolio B. Copeptin in the differential diagnosis of hyponatremia. J Clin Endocrinol Metab. 2009 Jan;94(1):123-9. doi: 10.1210/jc.2008-1426. Epub 2008 Nov 4. PMID 18984663
- [Background] Christ-Crain M, Morgenthaler NG, Fenske W. Copeptin as a biomarker and a diagnostic tool in the evaluation of patients with polyuria-polydipsia and hyponatremia. Best Pract Res Clin Endocrinol Metab. 2016 Mar;30(2):235-47. doi: 10.1016/j.beem.2016.02.003. Epub 2016 Feb 16. PMID 27156761
- [Background] Sailer CO, Winzeler B, Nigro N, Suter-Widmer I, Arici B, Bally M, Schuetz P, Mueller B, Christ-Crain M. Characteristics and outcomes of patients with profound hyponatraemia due to primary polydipsia. Clin Endocrinol (Oxf). 2017 Nov;87(5):492-499. doi: 10.1111/cen.13384. Epub 2017 Jul 7. PMID 28556237
- [Background] Boursier G, Almeras M, Buthiau D, Jugant S, Daubin D, Kuster N, Dupuy AM, Ribstein J, Klouche K, Cristol JP. CT-pro-AVP as a tool for assessment of intravascular volume depletion in severe hyponatremia. Clin Biochem. 2015 Jul;48(10-11):640-5. doi: 10.1016/j.clinbiochem.2015.03.013. Epub 2015 Mar 28. PMID 25828045
- [Background] Nigro N, Winzeler B, Suter-Widmer I, Schuetz P, Arici B, Bally M, Blum CA, Nickel CH, Bingisser R, Bock A, Huber A, Muller B, Christ-Crain M. Evaluation of copeptin and commonly used laboratory parameters for the differential diagnosis of profound hyponatraemia in hospitalized patients: 'The Co-MED Study'. Clin Endocrinol (Oxf). 2017 Mar;86(3):456-462. doi: 10.1111/cen.13243. Epub 2016 Oct 7. PMID 27658031
- [Background] Kumar S, Berl T. Sodium. Lancet. 1998 Jul 18;352(9123):220-8. doi: 10.1016/S0140-6736(97)12169-9. PMID 9683227